CLINICAL TRIAL: NCT01630395
Title: The Effect of Recruitment Maneuver With Protective Ventilation on the Pulmonary and Systemic Inflammatory Response to One-lung Ventilation
Brief Title: The Effect of Recruitment Maneuver With Protective Ventilation During Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JHBahk_recruitment maneuver
Record Dates: First submitted 2012-06-21; First posted 2012-06-28 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2012-06

CONDITIONS: Mechanical Ventilation Complication; Thoracic Surgery; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- conventional (No Intervention): Two-lung ventilation: tidal volume = 10 ml/kg, no PEEP. One-lung ventilation: tidal volume = 10 ml/kg, no PEEP
- Protective (Active Comparator): Two-lung ventilation: tidal volume 8 ml/kg, PEEP of 5 cmH2O. One-lung ventilation: tidal volume 6 ml/kg, PEEP of 5 cmH2O.
  Interventions: Procedure: protective ventilation
- Recruitment (Active Comparator): Two-lung ventilation: tidal volume 8 ml/kg, PEEP of 5 cmH2O. One-lung ventilation: tidal volume 6 ml/kg, PEEP of 5 cmH2O. Recruitment maneuver will be applied during one-lung ventilation.
  Interventions: Procedure: Recruitment maneuver combined with protective ventilation

INTERVENTIONS:
Procedure: protective ventilation — low tidal volume and PEEP
  Arms: Protective
Procedure: Recruitment maneuver combined with protective ventilation — Low tidal volume, PEEP and recruitment maneuver
  Arms: Recruitment

SUMMARY:
The purpose of this study is to determine if a recruitment maneuver combined with protective ventilatory strategy could reduce the pulmonary and systemic inflammatory responses to one-lung ventilation during thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* 20 Years and older
* Patients undergoing thoracic surgery

Exclusion Criteria:

* Emergency surgery
* Heart failure
* Pulmonary hypertension
* Forced vital capacity or forced expiratory volume in 1 sec < 50% of the predicted values
* Coagulation disorder
* Pulmonary or extrapulmonary infections
* History of treatment with steroid in 3 months before surgery
* History of recurrent pneumothorax
* History of lung resection surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Levels of IL-8, TNFa in the bronchoalveolar lavage | up to 20 minutes, after reexpansion of the non-dependent lung at the end of surgery

SECONDARY OUTCOMES:
Levels of IL-1, IL-6, IL-10 in the bronchoalveolar lavage | up to 20 minutes, after reexpansion of the non-dependent lung at the end of surgery
plasmatic concentration of inflammatory mediators IL-1, IL-6, IL-8, IL-10, TNFa | up to 20 minutes, after reexpansion of the non-dependent lung at the end of surgery
oxygenation | 1 hour after extubation
  Changes in PaO2/FIO2 ratio
Chest-X ray | 7 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea